CLINICAL TRIAL: NCT06153043
Title: Fertility and Pregnancy in Patients With Classic Congenital Adrenal Hyperplasia
Acronym: FERTI-HCS
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_1153; 2023-A02432-43 (Other: ID-RCB)
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Classic Congenital Adrenal Hyperplasia
Keywords: Classic congenital adrenal hyperplasia; fertility; fecundity; pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Women patients with classical congenital adrenal hyperplasia — The Easily and Médifirst medical files of these patients will be studied in order to collect the desired variables. If the files are incomplete, and if data concerning fertility, pregnancy, and the characteristics of the newborn are missing, patients will be contacted to ask them to answer the questionnaire to obtain this information.

SUMMARY:
Classic congenital adrenal hyperplasia (CAH) is a rare genetic endocrine disorder. Its prevalence is around 1/15.000. It results from a deficiency in 21-hydroxylase, an adrenal steroidogenic enzyme involved in the biosynthesis of cortisol and aldosterone. Enzyme deficiency in the steroideogenesis pathway leads to cortisol and aldosterone deficiency of varying severity, and to the accumulation of precursors (17OHP and Progesterone), which are diverted to the production of androgens (Testosterone and D4AD).

There are two clinical forms of classical CAH : the salt wasting form and the simple virilizing form, depending on the degree of aldosterone deficiency.

The clinical signs are adrenal insufficiency and hyperandrogenism. Hyperandrogenism manifests itself during foetal life, and may be responsible for virilization of the external genitalia of a female foetus, of varying severity.

The challenge in managing this condition is to find the right therapeutic balance. Hydrocortisone and fludrocortisone supplementation must be adapted to control adrenal insufficiency, and limit hyperandrogenism. It must be sufficient to avoid episodes of acute adrenal insufficiency, but not excessive to avoid complications secondary to hypercorticism.

During childhood, this balance is necessary for growth and pubertal development. However, this balance is difficult to achieve and maintain over time.

In adulthood, the fertility of patients is an important issue. This one remains poorly understood.

It was only after the introduction of cortisol supplementation in the treatment of CAH in the 1950s that the first pregnancies were described. Since when, due to the rarity of the pathology, the number of pregnancies studied has remained low, and the literature has little hindsight on the subject.

This pathology has long been associated with female infertility, due to many factors : biological, mechanical, psychological and sexual, among others. Biological hyperandrogenism may be responsible for chronic dysovulation, and may render the endometrium unsuitable for embryonic implantation. The virilization of the external genitalia and possible complications of pelvic surgery can be an obstacle to sexuality in these patients. They experience sexual difficulties, particularly during penetrative intercourse. The literature also shows that the majority of these patients are single and that their sexual orientation is more likely to be homosexual. Finally, the desire to have children is less prevalent in these patients than in the general population.

The first published studies on the fertility of CAH patients showed a lower pregnancy rate than the general population, but did not take into account the patient' desire to become pregnant.

In 2009, Casteras et al demonstrated for the first time in a cohort of CAH patients that fecundity is preserved in patients with a desire to become pregnant.

It should be noted that the fertility of patients with CAH may evolve in the coming years in France thanks to the new bioethics law voted in 2021, which now allows unmarried patients and patients in homosexual couples to have access to male gamete donation.

In addition, very little is known about the course of pregnancies in patients with CAH. Few pregnancies have been studied to date.

Hormonal balance during pregnancy if difficult to monitor, given the absence of reliable biological makers during this period. In this context, it is complicated to know the impact of the pathology and its balance on the course of the pregnancy.

The latest articles published on the subject of pregnancy complications are contradictory. Some find an increased risk of gestational diabetes. Others find a higher risk of maternal-fetal infection, low weight for gestational age, or congenital malformations than in general population. The increased risk of miscarriage is debated.

On the other hand, articles are unanimous on the most frequent mode of delivery in this population : in the vast majority of cases, patients give birth by ceasarian section, due to their history of pelvic surgery.

It is in context that we wish through this study to make a point of fertility and pregnancy in patients with classical CAH.

ELIGIBILITY:
Inclusion Criteria:

for patient :

* Adult patient > 18 years
* Classical congenital adrenal hyperplasia (21-hydroxylase deficiency, 11β-hydroxylase deficiency and 3βHSD2 deficiency)
* Who have indicated that they do not object to participating in the sudy

For partners :

- No objection to the collection of their fertility data

Exclusion Criteria:

* Non classical congenital adrenal hyperplasia
* Classical congenital adrenal hyperplasia due to other enzyme block

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will focus on patients in the Endocrinology department of the Louis Pradel Hospital in Bron, suffering from a classic form of Congenital Adrenal Hyperplasia by enzymatic block.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Describe the fertility of classical CAH women patients who had a desire for pregnancy and sought to conceive | At inclusion
  Proportion of patients who have had at least one pregnancy, regardless of outcome, among patients who have had a desire for pregnancy and have tried to conceived

CONTACTS AND LOCATIONS:
Locations (1):
- Endocrinology Department of Louis Pradel Hospital, Bron, France

IPD SHARING:
Plan to Share IPD: No